CLINICAL TRIAL: NCT05742711
Title: Efficacy of Percutaneous Electrical Neurostimulation (PENS)of the Auricle as an Opioid Sparing Postoperative Analgesic Technique in Cancer Endometrium and Cancer Cervix
Brief Title: Efficacy of PENS of the Auricle as an Opioid Sparing Postoperative Analgesic Technique in Cancer Endometrium and Cancer Cervix Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DyAnsys, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CS015
Record Dates: First submitted 2023-02-02; First posted 2023-02-24 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Cancer of Endometrium; Cancer of Cervix
MeSH Terms: conditions — Endometrial Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): The group who have received PENS treatment using PrimaryRelief in addition to Injection paracetamol in a dosage of 15mg/kg every 6th hourly. Break through pain with NRS>4 will be managed with injection tramadol at 1mg/kg followed by 0.5mg/kg after 10mins in cases of persisting pain.
  Interventions: Device: Primary Relief
- Control Group (Sham Comparator): The group who have received a sham device along with Injection paracetamol in a dosage of 15mg/kg every 6th hourly. Break through pain with NRS>4 will be managed with injection tramadol at 1mg/kg followed by 0.5mg/kg after 10mins in cases of persisting pain.
  Interventions: Device: Primary Relief - Sham Device

INTERVENTIONS:
Device: Primary Relief — Continuous neurostimulation with a set of pre-assigned stimulation parameters.
  Other Names: Percutaneous Electrical Nerve Stimulator (PENS)
  Arms: Treatment Group
Device: Primary Relief - Sham Device — Standard treatment with the application of sham device shall be followed with additional analgesics available if necessary.
  Other Names: Standard Treatment for Postoperative Pain
  Arms: Control Group

SUMMARY:
Pain relief following laparotomy surgery requires a variety of techniques including invasive ones like epidural or nerve blocks along with different classes of drugs, out of which opioids are most predominant. Each of these drugs have with their own set of advantages and also side effects. An ideal common system of analgesia is not possible due to patient variability. And no drug is devoid of side effects. Hence the aim is to ensure effective analgesia using drugs or techniques which are minimally invasive with negligible side effects.

DETAILED DESCRIPTION:
Efficient post operative pain relief is an essential part of comprehensive recovery of patients. Conventional method of pain management of laparotomy surgeries in CA endometrium and cervix patients involves invasive techniques like epidural or selective nerve block coupled with a varied choice of analgesics like opioids, NSAID or acetaminophen, wherein each drug is associated with its own set of contraindications and side effects. Despite advances in analgesic regimen including multimodal analgesic regimen, opioids have been observed to remain the mainstay postoperative analgesia in cancer patients despite its well-established side effects.

This double-blinded prospective interventional study is conducted to explore the alternative of percutaneous electrical nerve stimulation (PENS) devices for effective pain relief with minimal to no side-effects.

The device will have tiny needles and a battery system that will be placed on and behind the patient's ear when they are under anesthesia.

It acts by stimulating nerves around ear region by series of pain free impulse generation leading to centrally (brain) mediated response by altering certain chemical substances responsible for causing pain thereby providing relief for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 yrs
* Diagnosed with CA-endometrium OR CA -cervix of stage I/II and post RT CA cervix patients coming for hysterectomy
* Elective surgery
* Informed consent obtained
* ASA (American Society of Anaesthesiology) physical status 1-3

Exclusion Criteria:

* Patient refusal
* Cancer cervix other than the stages mentioned in inclusion criteria ASA PS >3
* Emergency surgery, Laparoscopic and robotic procedures
* Unplanned postoperative ventilation
* Allergy/sensitivity to adhesive
* Active skin infection/lesion in the ear region
* H/O of seizure or cerebral disease
* H/O chronic pain and prolonged analgesic usage
* H/O opioid dependence
* H/O anxiety or psychiatric illness requiring treatment
* Pre-existing implantable/ electronic on demand device
* Patients who might require MRI in the study period
* Patients with transmissible diseases
* Patients with coagulopathies
* Absolute or relative contraindication to drugs used in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-05-16 (Actual); Primary Completion 2025-01-13 (Actual); Study Completion 2025-01-13 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale (NRS) | 0 - 4 days; 0 hours, 2 hours, 4 hours, 8 hours, 12 hours, 18 hours, 24 hours, 36 hours, 48 hours, 72 hours, 96 hours. Outcomes will be reported as an average over each individual postoperative day and as an average over 5 days independently for rest.
  The primary goal is to evaluate the efficacy of PENS treatment in the change in postoperative pain after cancer surgery compared to the control group. The pain is measured using the numerical rating scale (NRS). Pain Score will be measured on a scale (0 = no pain;10 = worst imaginable pain; lower scores indicate better outcome)

SECONDARY OUTCOMES:
Overall Postoperative analgesia and opioid requirement | 0 - 4 days, duration and dose of all prescriptions are recorded.
  To evaluate the effect of treatment in reducing the overall postoperative analgesia and opioid requirement. We will record the total dose and duration of additional analgesics required from the immediate postoperative period till pod 4 in iv morphine equivalents.
Patient Ambulation | 1 - 4 days; 24 hours, 36 hours, 48 hours, 72 hours, 96 hours.
  Evaluate the ease of patient ambulation by assessing associated Numeric Rating Scale (NRS) score (0 = no pain;10 = worst imaginable pain; lower scores indicate better outcome)
Record of Participant Bowel Movement Patterns | 0 - 4 days; Whenever the patient experiences the bowel movement.
  Onset of Bowel Movements - POD 1/POD 2/ POD 3/ > POD3
Richmond Agitation Sedation Scale (RASS) | 0 - 4 days; 0 hours, 2 hours, 4 hours, 8 hours, 12 hours, 18 hours, 24 hours, 36 hours, 48 hours, 72 hours, 96 hours.
  Compare Richmond Agitation Sedation Scale (RASS) score at a different time point during the follow-up time. RASS score will be measured on a scale (from -5 = Unarousable to +4 = Combative where 0 = Alert and calm)
Patient Discomfort | Time Frame: 0 - 4 days; Whenever the patient experiences the discomfort.
  Patient Discomfort due to device (Yes / no)
Bleeding | Time Frame: 0 - 4 days; Whenever the patient experiences bleeding.
  Bleeding at the site of device placement (Yes / No)
Interference with Daily Activities | Time Frame: 0 - 4 days; Whenever the patient experiences disruption in daily activities.
  Interference with activities of daily living due to the device (Yes/No)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Sahithya Sriman, MBBS, MD, Principal Investigator — Cancer Institue, WIA,
Locations (1):
- Cancer Institute,(Wia), Chennai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Arponrat P, Pongrojpaw D, Tanprasertkul C, Suwannarurk K, Bhamarapravatana K. Postoperative Pain Relief in Major Gynaecological Surgery by Perioperative Parecoxib Administration: Thammasat University Hospital Study. J Med Assoc Thai. 2015 Jul;98(7):636-42. PMID 26267984
- [Result] Pogatzki-Zahn E, Kutschar P, Nestler N, Osterbrink J. A Prospective Multicentre Study to Improve Postoperative Pain: Identification of Potentialities and Problems. PLoS One. 2015 Nov 24;10(11):e0143508. doi: 10.1371/journal.pone.0143508. eCollection 2015. PMID 26600464
- See also: Pattern of use of analgesics in post-operative pain management in adults undergoing laparotomy surgery: a prospective observational study — https://www.ijsurgery.com/index.php/isj/article/view/2388